CLINICAL TRIAL: NCT03921827
Title: External Counterpulsation Therapy for Symptomatic and Severe Steno-occlusive Disease of Intracranial Internal Carotid or Middle Cerebral Artery and Impaired Cerebral Vasodilatory Reserve
Brief Title: External Counterpulsation Therapy for Severe Steno-occlusive Intracranial Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, VIJAY KUMAR SHARMA, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUSingapore_EECP
Record Dates: First submitted 2019-04-14; First posted 2019-04-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
Keywords: MCA; ICA; vasodilatory reserve; EECP; intracranial stenosis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 1:1 allocation to EECP therapy and best medical therapy
Who Masked: Outcomes Assessor
Masking Description: Outcome will be assessed by independent assessors for stroke/TIA recurrence within 6 months as well as change in cerebral vasodilatory reserve on acetazolamide challenged HMPAO- SPECT of brain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EECP therapy (Experimental): Half of the study sample will be allocated to EECP therapy (35 sessions) of 1-hour each. Acetazolamide challenged HMPAO-SPECT will be performed before randomization and repeated 2-months after the completion of EECP therapy. MRI of the brain would be performed after completion of EECP therapy to document any silent stroke.
  Interventions: Device: Enhance External Counterpulsation Therapy
- Best Medical Therapy (No Intervention): This group will receive the best medical therapy according to our institutional practice and as per the recommendations of American Stroke Association.

INTERVENTIONS:
Device: Enhance External Counterpulsation Therapy — EECP therapy would be administered to this group for 1-hour a day for a total of 35 sessions
  Arms: EECP therapy

SUMMARY:
Intracranial stenosis is prevalent among Asians and constitute a common cause of cerebral ischemia. While the best medical therapy carries stroke recurrence rates in access of 10% per year, intracranial stenting was associated with unacceptable peri-procedural ischemic events. Cerebral ischemic events are strongly related to the severity of intracranial stenosis, being high in patients with severe intracranial stenosis with poor vasodilatory reserve. Enhanced External Counter-Pulsation (EECP) therapy is known to improve myocardial perfusion by facilitating the development of collateral blood vessels in the heart. The investigators hypothesize that EECP therapy may be useful in patients with severe stenosis of intracranial internal carotid (ICA) or middle cerebral artery (MCA).

DETAILED DESCRIPTION:
Among Asian patients, intracranial stenosis is more common and accounts for about 30-50% of all strokes. The risk of recurrent stroke or TIA in presence of intracranial stenosis of a major intracranial artery and recent TIA/ stroke is about 23% at 1 year despite treatment. Recurrence rate for stroke/TIA in intracranial atherosclerosis is dependent on degree of stenosis as well as presence of collaterals. In WASID study, patients with more than 70% stenosis had greater risk of recurrent event then those with 50-69%. Interestingly, patients with more than 70% intracranial stenosis with good collaterals demonstrated a lower risk for subsequent cerebral ischemic events.

The two main mechanisms of ischemic stroke (IS) in these patients are thromboembolism and cerebral hemodynamic insufficiency. While Transcranial Doppler (TCD) monitoring can establish thrombo-embolic phenomenon and help in planning the appropriate antithrombotic treatment, assessment of dynamic cerebral hemodynamic insufficiency remains a complex issue, and may serve as a potential target for improving the outcomes (and reducing recurrent cerebral ischemia) in patients with severe intracranial stenoses.

Treatment options for Intracranial stenosis:

Anti-platelet agents are recommended for secondary prevention of IS. WASID trial compared warfarin with INR of 2-3 against aspirin, did not show any difference in outcome of stroke recurrence. Furthermore, aspirin was found to be safer as compared to warfarin.

Use of short-term double antiplatelet therapy is shown to be effective in reducing stroke/TIA recurrence risk. In CLAIR study, patients with recent symptoms (</=7 days) and with intracranial stenosis were randomized to clopidogrel and aspirin versus aspirin monotherapy. Combination anti-platelet therapy reduced micro-embolic signals on TCD on Day 2 and 7. Use of double antiplatelet in intracranial stenosis was also supported by findings of SAMMPRIS trial in which patient with recent stroke of TIA with 70-99% intracranial stenosis were randomized to angioplasty or maximal medical treatment. The 90 day recurrence risk of 5.8% in the medical arm was much lower than 10.7% recurrence rate observed in WASID trial.

Surgical treatment:

Extracranial to intracranial bypass has been compared with medical management in patients with intracranial stenosis and it did not lower the risk of recurrent ischemic stroke. Furthermore, it was associated with worse outcome as compared to medical management. Also, the recently published COSS study failed to show any benefit of surgical treatment for carotid occlusion, largely related to better than expected event rates in the medical arm.

Endovascular Treatment:

Endovascular treatment has been used as a potential therapeutic option for intracranial atherosclerosis. In 2005, FDA approved self expanding Wingspan stent for use in medically refractory patients who harbor 50-99% stenosis of major intracranial artery. In 2011 Chimowitz et al published results of SAMMPRIS trial, which compared percutaneous trans-luminal angioplasty and stenting with medical management. Patients with recent TIA or stroke attributed to 70-99% stenosis of intracranial vessels were recruited in this trial. Enrollment of this trial was stopped after 451 patients were recruited as angioplasty and stenting group was associated with 14.7% event rate (stroke or death) at 30-days as compared to medical management arm (5.8% event rate).

Cerebral vasodilatory reserve:

The assessment of cerebral vasodilatory reserve (CVR) in patients with persistent arterial occlusive disease is important since inadequate CVR in symptomatic patients is considered a major risk factor for subsequent ischemic events. By using refined techniques for measuring cerebral blood volume (CBV) and cerebral blood flow (CBF), in addition to standard clinical and angiographic studies, it is possible to identify a small subgroup of patients with impaired CVR who are at risk of subsequent stroke. Accordingly, impaired CVR is often regarded as the basis for performing extra-/intracranial (EC/IC) bypass surgery with the aim of increasing CBF and restore CVR in this highly selected patient subgroup.

Identifying patients who are at increased risk for hemodynamic stroke is important because they may benefit from flow augmentation procedures, such as carotid endarterectomy, EC-IC bypass, or even angioplasty. The cerebral hemodynamic status can be determined by measuring CBF before and after vasodilatory challenge, which can be done with either hypercapnia or acetazolamide. Acetazolamide, a carbonic anhydrase inhibitor, has been shown to increase CBF in healthy subjects by inducing transient vasodilatation.

Cerebral autoregulation enables a constant CBF over a wide range of systemic blood pressure by varying the diameter of the intracranial arterioles. This may fail in some patients with severe steno-occlusive disease. TCD can measure vasomotor reactivity (VMR) by assessment of flow velocities in response to increasing carbon dioxide levels. This can be performed by simple breath-holding test and calculating the so-called 'breath holding index (BHI)', BHI is calculated as the relative increase in the MFV during breath holding divided by the time of apnea in seconds. In normal persons, the BHI amounts to 1.2±0.6. Silverstrini et al prospectively evaluated BHI in case-controlled studies and showed that impaired VMR can help to identify patients at higher risk of stroke in a population with asymptomatic carotid stenosis or a previously symptomatic carotid occlusion. A decreased VMR suggests failure of collateral flow to adapt to the stenosis progression. Various studies, using different provocative measures for assessing the VMR, demonstrated a remarkable ipsilateral event rate of around 30% (30% risk of stroke/ TIA during about 2 years).

In a recent study, the investigators demonstrated the phenomenon of 'intracranial steal' in patients with persisting intracranial occlusions where, hypercapnia can paradoxically decrease the residual flow velocity in the affected vessel at the expected time of normal brain vasodilation when blood pool is shifted to non-ischemic areas. The phenomenon of "reversed Robin Hood", an analogy with "rob the poor to feed the rich" was replicated by acetazolamide-challenged HMPAO-SPECT imaging. The investigators have demonstrated recently the value of multimodality evaluation of CVR is feasible and may aid in taking therapeutic decisions regarding revascularization procedures.

Enhanced External Counter Pulsation (EECP) is a new noninvasive therapy used to treat patients with angina, congestive heart failure, acute myocardial infarction and cardiogenic shock by augmenting blood flow to the cardiac and systemic arterial circuits. EECP's hemodynamic effects include 20% to 25% improvement in arterial flow volume in the carotid, renal and hepatic arteries, with a 20% to 40% improvement in coronary artery blood flow accompanied by a 12% increase in left ventricular (LV) stroke volume.

EECP as a frontline treatment for revascularization in patients with angina refractory to medical therapy has shown similar findings to coronary artery bypass and percutaneous coronary interventions including improvement in cardiac functional class, decreased anginal episodes, and reduction in nitroglycerin use. EECP has been shown to produce similar hemodynamic effects to intra-aortic balloon pumps (IABP), yet is a noninvasive technology carrying less implementation risk.

Lastly, TCD measurements in recovering ischemic stroke patients undergoing EECP have demonstrated a significant increase in MCA flow velocities. Peak diastolic augmented velocities (PDAV) averaged 72 + 29 cm/second a 196% increase in flow(RMCA), and 78 + 30 cm/second a 199% increase in flow (LMCA) on EECP, significantly higher than pre-procedural EDV (RMCA 37+11cm/second, p=0.014; LMCA 39+9cm/second, p=0.022). Given the altered waveform morphology, traditional calculation of MFV using peak systole and end-diastole would fail to capture EECP's flow augmentation effects. Augmented MFV (AMFV) was recalculated by substituting EDV with a measure derived from the summed average of PDAV and EDV (augmented diastolic velocity [ADV]).

Patients in whom a long stenotic segment involved both terminal ICA and proximal MCA would be classified as having a steno-occlusive disease of terminal ICA. Steno-occlusive disease of ICA or MCA would be considered severe (>70%) according to the velocity criteria and presence of 'blunted' flow spectra in the arterial segment distal to the stenosis. Therefore, tandem lesions in a single arterial tree (intracranial ICA and MCA, proximal MCA and distal MCA, extracranial ICA and ipsilateral intracranial ICA or extracranial ICA and ipsilateral MCA), if associated with blunted flow spectra in distal MCA would qualify the criteria for >70% stenosis. Importantly, the TCD diagnostic criteria for intracranial stenosis in our neurovascular laboratory have been validated against CT angiography.

Patients would be randomized (1:1 by using drawing previously prepared chits in a bag) into either maximal medical management (plus sham EECP) or maximal medical management plus EECP. EECP sessions are planned 5 times/week for a total of 35 sessions. CVR would be measured at baseline as well as at 4 months of EECP treatment initiation. Improvement in CVR on symptomatic side would be measured by TCD-BHI as well as acetazolamide challenged HMPAO-SPECT and compared with patients in medical management (and sham EECP) arm for significant difference. Patients will also be followed up for recurrence of stroke/TIA during the study period.

Maximal medical management would be same in both groups as per the current AHA/ASA guidelines. Briefly, all ischemic stroke cases with intracranial stenosis receive dual antiplatelet agents (aspirin and clopidogrel for 1 month followed by clopidogrel or aspirin long term). The investigators aim to keep HbA1c at 7% or less in all cases. Blood pressure target in the stroke patients eligible for this study (at least 1 month after acute stroke) is less than 140/90mmHg. For lipids, the target LDL is less than 2.6mmol/L.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recent stroke/TIA and severe stenosis of intracranial ICA or MCA and impaired CVR within previous three months but not before 3 weeks after acute stroke. This is to differentiate between patients with a long-standing fixed-stenosis from patients with partially recanalized intracranial artery (masquerading as severe stenosis).
2. Age >21 years

Exclusion Criteria:

1. Patients with atrial fibrillation/ arrhythmias.
2. Within 2 weeks of cardiac catheterization or arterial puncture at femoral puncture site.
3. Decompensated heart failure , usually class 3 or 4
4. LV EF <30%
5. Moderate or severe AR
6. Persistent and uncontrolled hypertension (BP persistently >160/100 mmHg)
7. Bleeding diathesis
8. Active thrombophlebitis/ venous disease of lower limbs
9. Severe lower extremity vaso-occlusive disease
10. Presence of a documented aortic aneurysm/ dissection requiring surgical repair
11. Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Improvement in cerebral vasodilatory reserve | at baseline and after 2 months of the completion of EECP therapy
  To evaluate whether Enhanced External Counter-Pulsation (EECP) therapy would lead to a change in cerebral vasodilatory reserve (CVR) by at least 4% in patients with severe and recently symptomatic stenosis of intracranial carotid (ICA) or middle cerebral artery (MCA).

SECONDARY OUTCOMES:
Stroke TIA/recurrence | at 6 months
  To evaluate the impact of EECP on recurrence of cerebral ischemic event in patients with severe and recently symptomatic stenosis of ICA or MCA.
Impact of EECP on cognition | at 6 months
  To evaluate the impact of EECP on change in neurocognitive performance by at least 2 points (60 minutes protocol suggested by NINDS harmonization workshop) in patients with severe and recently symptomatic stenosis of ICA or MCA.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay K Sharma, MD, Principal Investigator — National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, the team would be happy to share the anonymised database to any study with a similar protocol
Supporting Information: Study Protocol, CSR
Time Frame: After completion of the study
Access Criteria: The data will be shared via email to the PIs of studies with a similar protocol

REFERENCES:
- [Derived] Sharma VK, Gopinathan A, Tan BYQ, Loh PH, Hung J, Tang D, Chua C, Chan ACY, Ong JJY, Chin A, Jing M, Goh Y, Sunny S, Keat CH, Ka Z, Pandya S, Wong LYH, Chen JT, Yeo LLL, Chan BPL, Teoh HL, Sinha AK. Enhanced external counter pulsation therapy in patients with symptomatic and severe intracranial steno-occlusive disease: a randomized clinical trial protocol. Front Neurol. 2023 May 30;14:1177500. doi: 10.3389/fneur.2023.1177500. eCollection 2023. PMID 37325226